CLINICAL TRIAL: NCT00499356
Title: Shear and Pressure Reducing Insoles for the Diabetic Foot
Acronym: GlideSoft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetica Solutions Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DK55909
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2007-07-11 (Estimated); Status verified 2007-07

CONDITIONS: Diabetes; Ulceration; Amputation; Foot Deformity; Neuropathy
Keywords: friction; pressure; insole; ulcer; prevention
MeSH Terms: conditions — Diabetes Mellitus; Ulcer; Foot Deformities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: pressure reducing insole
Device: GlideSoft®

SUMMARY:
We evaluated the feasibility of the GlideSoft™ novel insole to reduce pressure and shear forces on the foot. No commercially available insoles are designed to reduce shear. Although insurance providers spend millions on diabetics' therapeutic insoles, there is no scientific data about shear or pressure reduction. We will evaluate the optimal bonded materials from Phase I compared to the Glidesoft™ design using the same combination of viscoelastic materials. We evaluate 2 patient groups of 150 patients per arm (300 total) in an 18 month trial. The control group patient arm wore a traditional bonded insole whereas another the second arm receive the GlideSoft™. At baseline, and at the end of the 18 month trial, in-shoe gait lab and in vitro biomechanical parameters measured pressure, shear, and material properties as these changed with wear. This Phase II eighteen (18) month clinical trial evaluated the effectiveness of ShearSole™ reducing the incidence of diabetic ulcers. The overall study hypothesis was that GlideSoft™ provides significant shear reduction as compared to traditional insoles without sacrificing pressure reduction characteristics or durability.

DETAILED DESCRIPTION:
1. To evaluate the efficacy of a shear reducing shoe insole (GlideSoft) in reducing the incidence of diabetic foot pathology among high-risk patients. We studied the effectiveness of a shear reducing shoe insole to prevent foot ulcers in high-risk diabetics with sensory neuropathy, a history of a foot ulcer or a history of a partial foot amputation. The study comprised two treatment arms. The first group received standard therapy involving standard therapeutic shoes and insoles, patient education and regular foot evaluations by a physician. The second group received the same standard therapy, but instead of the standard insoles patients used the GlideSoft - a novel shear reducing insole. As determined in the Phase I study, the GlideSoft dramatically reduced shear forces compared to standard insoles, while performing equally well in reducing compressive forces. Patients were followed for 18 months. The primary study outcome was for incident foot ulcers. Our hypothesis was that patients who use the GlideSoft will have fewer ulcers and that these ulcers will be less severe compared to patients evaluated in the Standard Insole Group.
2. To evaluate changes in pressure and shear reducing capabilities of the two. To evaluate changes in pressure and shear reducing capabilities of the GlideSoft and standard insoles over the duration of use.

   We measured in-shoe pressures and in-vitro shear forces at the foot-insole interface at the beginning of the study and after patients wore the insole for four months or one "standard cycle of wear". We used the Novel Electronics, Inc. Pedar in-shoe pressure system to measure the interface between the foot and insole and the Shear Force Tester (see Phase I report) to evaluate shear forces. We expected that the GlideSoft would significantly reduce shear forces and provide equivalent reduction in vertical forces at both the day 0 evaluation and day 120 evaluations.
3. To evaluate patient perceived benefits, satisfaction, and compliance with the 2. To evaluate changes in pressure and shear reducing capabilities of the GlideSoft and standard insoles over the duration of use.

We measured in-shoe pressures and in-vitro shear forces at the foot-insole interface at the beginning of the study and after patients wore the insole for four months or one "standard cycle of wear". We used the Novel Electronics, Inc. Pedar in-shoe pressure system to measure the interface between the foot and insole and the Shear Force Tester (see Phase I report) to evaluate shear forces. We expected that the GlideSoft would significantly reduce shear forces and provide equivalent reduction in vertical forces at both the day 0 evaluation and day 120 evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes by WHO criteria
* Ability to provide informed consent
* 18-80 years of age

Exclusion Criteria:

* Patients with open ulcers or open amputation sites
* Active Charcot arthropathy
* Severe peripheral vascular disease
* Active foot infection
* Dementia
* Impaired cognitive function
* History of drug or alcohol abuse within one year of the study
* Other conditions based on the PI's clinical judgment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2002-05; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Incident foot ulcers | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin R Higgins, DPM, Principal Investigator
Locations (1):
- Kevin R. Higgins, DPM, San Antonio, Texas, United States

REFERENCES:
- [Result] Lavery LA, Higgins KR, Lanctot DR, Constantinides GP, Zamorano RG, Athanasiou KA, Armstrong DG, Agrawal CM. Preventing diabetic foot ulcer recurrence in high-risk patients: use of temperature monitoring as a self-assessment tool. Diabetes Care. 2007 Jan;30(1):14-20. doi: 10.2337/dc06-1600. PMID 17192326
- [Derived] Lavery LA, LaFontaine J, Higgins KR, Lanctot DR, Constantinides G. Shear-reducing insoles to prevent foot ulceration in high-risk diabetic patients. Adv Skin Wound Care. 2012 Nov;25(11):519-24; quiz 525-6. doi: 10.1097/01.ASW.0000422625.17407.93. PMID 23080240